CLINICAL TRIAL: NCT02959697
Title: Subconjunctival Injection of Local Anesthetic in Anterior Blepharoptosis Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: HS20066 (B2016:085)
Record Dates: First submitted 2016-10-31; First posted 2016-11-09 (Estimated); Last update posted 2022-06-10 (Actual); Status verified 2022-05

CONDITIONS: Blepharoptosis; Ptosis
Keywords: Blepharoptosis; Ptosis; Surgery; Pain Reduction; Anesthetic; Local Anesthetic; Subconjunctival
MeSH Terms: conditions — Blepharoptosis | interventions — Lidocaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subcut. + Subconj. Injection (Experimental): Patients will undergo standard blepharoptosis repair using an anterior approach, with an added injection of local anesthetic (Xylocaine) beneath the conjunctiva of the lid being operated on. They will still receive the standard subcutaneous local anesthetic given during blepharoptosis repair.
  Interventions: Drug: Subcut. + Subconj. Xylocaine; Procedure: Blepharoptosis Repair
- Subcut. + Sham Subconj. Injection (Sham Comparator): Patients will undergo standard blepharoptosis repair using an anterior approach, however they will not receive the additional subconjunctival Xylocaine injection. Instead, they will receive a sham injection of Normal Saline to prevent them from knowing which eye received the additional anesthetic.
  Interventions: Drug: Subcut. + Sham Subconj. Injection; Procedure: Blepharoptosis Repair

INTERVENTIONS:
Drug: Subcut. + Subconj. Xylocaine — Patient will receive the standard subcutaneous local anesthetic as well as an additional subconjunctival injection of local anesthetic (Xylocaine).
  Other Names: Xylocaine
  Arms: Subcut. + Subconj. Injection
Drug: Subcut. + Sham Subconj. Injection — Patient will receive the standard subcutaneous local anesthetic as well as a subconjunctival sham injection of Normal Saline.
  Other Names: Normal Saline
  Arms: Subcut. + Sham Subconj. Injection
Procedure: Blepharoptosis Repair — Patients will undergo blepharoptosis repair using an anterior approach.
  Other Names: Ptosis Repair

SUMMARY:
Blepharoptosis (ptosis) repair is a common and generally well tolerated surgical procedure usually performed using local anesthetic. However, a subset of patients appears to experience intraoperative pain/discomfort during ptosis repair using an anterior approach with subcutaneous local anesthetic. Posterior subconjuctival local anesthetic is currently used for eyelid procedures such as chalazion incision and drainage and full-thickness eyelid resections. The purpose of this study is to determine whether an additional subconjunctival injection of local anesthetic, through the posterior aspect of the eyelid, reduces intraoperative pain during anterior ptosis repair.

DETAILED DESCRIPTION:
Patients will be recruited from Dr. Matthew Lee-Wing's practice. Eligible participants include those requiring bilateral blepharoptosis repair requiring an anterior surgical approach. The patient will need to have a similar degree of ptosis in each eye (as measured by each eye's "Marginal Reflex Distance #1"). Patients will be given information regarding the outcomes of interest, and informed re: risks and benefits of participating.

Upon agreeing to participate, the patient will be asked to sign a consent form indicating their wish to participate in the study (see below).

Each patient will have blepharoptosis repair surgery on both of their eyes. One eye will act as a control in that the operation will proceed in a manner in-line with current practice (IE with subcutaneous local anesthetic alone). The other eye will receive both subcutaneous local anesthetic, as well as an additional injection of local anesthetic underneath the conjunctiva of the upper eyelid (IE on the inner surface of the eyelid). The eye/side receiving only the standard, subcutaneous local anesthetic will also receive a sham injection of normal saline in order to prevent the patient from knowing which side is receiving the additional anesthetic dose. Dr. Lee-Wing will perform all of the surgeries within the study, and will be blinded as to which patient is receiving the additional anesthetic. The blinding will be accomplished by the assisting treatment room nurse, who will use an algorithm to randomly select which eyelid will receive the subconjunctival Xylocaine and which will receive the subconjunctival Normal Saline.

Following their procedure, each patient will complete a questionnaire designed to assess their intraoperative pain.

Statistical analysis will be performed, and will compare the patient's intraoperative pain rating for the eyelid that received the sham Normal Saline injection and the eyelid that received the Xylocaine injection. The presence of post-operative lagophthalmos/fluorescein staining will be compared between the two groups, as will the post-operative Marginal Reflex Distance 1. The above comparisons will be made using McNemar's test.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years of age or older and able to give informed consent in English
* Must have bilateral blepharoptosis undergoing repair using an anterior approach
* The degree of ptosis must be approximately symmetrical, with a difference in margin-reflex distance of 1 mm or less between the two sides

Exclusion Criteria:

* Previous eyelid surgery or trauma
* Congenital, mechanical, myogenic or neurogenic forms of ptosis
* Unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
0-10 Numerical Pain Scale | 6 Years
  Patients will be asked to describe the intraoperative pain they experienced in each eye during surgery. Results will be compared with McNemar's test.

SECONDARY OUTCOMES:
Presence of post-operative lagophthalmos/fluorescein staining | 6 Years
  The presence or absence of lagophthalmos and fluorescein staining will be assessed in each eye at the post-operative follow up appointment, and will be compared with McNemar's test.
Post-Operative margin-reflex distance 1 | 6 Years
  Post-operative margin-reflex distance 1 (MDR1 - distance between the pupillary light reflex and the lower edge of the upper lid) will be measured in each eye. The difference between the MDR1 of each eye will be analyzed using paired Student's T-testing.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Lee-Wing, MD, Principal Investigator — University of Manitoba
Locations (2):
- Canada (2):
  - Buhler Eye Centre, Misericordia Hospital, Winnipeg, Manitoba
  - Private Office (Dr. Lee-Wing). 1010-233 Kennedy st., Winnipeg, Manitoba

DOCUMENTS (1):
  • Study Protocol (2022-06-06): https://cdn.clinicaltrials.gov/large-docs/97/NCT02959697/Prot_003.pdf